CLINICAL TRIAL: NCT01096550
Title: Intensive Outpatient v. Outpatient Treatment With Buprenorphine Among African Americans
Brief Title: Intensive Outpatient Versus Outpatient Treatment With Buprenorphine Among African Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Friends Research Institute, Inc. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1RC1DA028407-01 (NIH); 1RC1DA028407-01 (NIH)
Record Dates: First submitted 2010-03-30; First posted 2010-03-31 (Estimated); Results first posted 2013-10-17 (Estimated); Last update posted 2020-04-08 (Actual); Status verified 2020-03

CONDITIONS: Drug Dependence
Keywords: opioid dependence; outpatient treatment; intensive outpatient treatment
MeSH Terms: conditions — Substance-Related Disorders; Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive Outpatient (Experimental): Buprenorphine patients receiving 9 or more hours of outpatient counseling.
  Interventions: Behavioral: Intensive Outpatient
- Outpatient (Active Comparator): Buprenorphine patients receiving between 2 and 8 hours of outpatient counseling.
  Interventions: Behavioral: Outpatient

INTERVENTIONS:
Behavioral: Outpatient — Buprenorphine patients receiving 2 to 8 hours of outpatient counseling.
  Arms: Outpatient
Behavioral: Intensive Outpatient — Buprenorphine patients receiving 9 or more hours of outpatient counseling.
  Arms: Intensive Outpatient

SUMMARY:
The purpose of this study is to compare the effectiveness of different levels of counseling (intensive outpatient versus standard outpatient) on treatment outcomes for African American adult patients receiving buprenorphine in 2 formerly "drug-free" programs.

DETAILED DESCRIPTION:
This two-group randomized clinical trial will test the effectiveness of intensive outpatient (IOP) v. standard outpatient (OP) treatment in 272 heroin-dependent African American adults receiving buprenorphine in 2 formerly "drug-free" programs. Participants will be randomly assigned to one of the two treatment intensity conditions at intake and assessed at baseline, 3-, and 6-months post-baseline to determine treatment retention, frequency and severity of heroin and cocaine use, self-reported HIV-risk, quality of life, and to determine DSM-IV criteria for Full or Partial Remission of Opioid Dependence. Furthermore, patient factors potentially critical for treatment success (e.g., attitudes towards buprenorphine and average buprenorphine dose while in treatment) will be examined to determine their importance in influencing treatment outcomes. Moreover, both patient and staff attitudes and average buprenorphine dose will be evaluated to determine their respective relationships to treatment experiences and treatment retention.

ELIGIBILITY:
Inclusion Criteria:

* heroin-dependent adults
* new admissions to buprenorphine outpatient treatment

Exclusion Criteria:

* pregnancy
* acute medical or psychiatric illness

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2010-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shannon G Mitchell, PhD, Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Friends Research Institute, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: New patients entering buprenorphine treatment at one of the two participating outpatient "drug-free" treatment programs were block randomized to either intensive outpatient treatment (IOP) or standard outpatient treatment (OP). The study initially included a third clinic site, which was dropped due to insufficient enrollment at that site.
Pre-assignment Details: 345 patients were randomized. Of those, the following participants were excluded from the study shortly after random assignment: 21 were from the discontinued site, 2 were dropped because of non-standard clinic treatment track, 1 voluntarily withdrew, 2 were erroneously re-enrolled. We also excluded 19 non-African Americans, per study protocol.
Groups:
- Intensive Outpatient: Buprenorphine patients receiving 9 or more hours of outpatient counseling.
  Intensive Outpatient : Buprenorphine patients receiving 9 or more hours of outpatient counseling.
- Outpatient: Buprenorphine patients receiving between 2 and 8 hours of outpatient counseling.
  Outpatient : Buprenorphine patients receiving 2 to 8 hours of outpatient counseling.
Period: Overall Study
Arm/Group | Intensive Outpatient | Outpatient
Started | 170 | 175
Completed | 133 | 146
Not Completed | 37 | 29
Not completed — discontinued site | 10 | 11
Not completed — non-regular treatment track at clinic | 1 | 1
Not completed — clinic readmission | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — non-African American participant | 13 | 6
Not completed — Lost to Follow-up | 12 | 9

BASELINE CHARACTERISTICS:
Population: 21 were from the discontinued site, 2 dropped because participant was non-regular treatment track, 1 voluntarily withdrew from the study, 1 was erroneously re-enrolled after being re-admitted to the same clinic, and 1 was erroneously re-enrolled, and 19 were not African American.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensive Outpatient | Outpatient | Total
Number analyzed (Participants) | 170 | 175 | 345
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 168 | 174 | 342
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.15 (8.15) | 46.27 (6.75) | 45.23 (7.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 67 | 129
  Male | 108 | 108 | 216
Region of Enrollment [Number; unit: participants]
  United States | 170 | 175 | 345

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Meeting Diagnosis of Opioid Dependence on Composite International Diagnostic Interview-2 (CIDI-2)
Time Frame: 6 months post-baseline
Measure: Number; unit: percentage of opioid dependent subjects
Arm/Group | Intensive Outpatient | Outpatient
Number analyzed (Participants) | 145 | 155
percentage of opioid dependent subjects | 20 | 21

ADVERSE EVENTS:
Description: serious and/or other [non-serious] adverse events were not collected/assessed
Arm/Group | Intensive Outpatient | Outpatient
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
OP condition participants received more counseling services at the clinics as part of their regular care than was initially expected and IOP condition participants received slightly less that 9 hours of counseling, on average.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No